CLINICAL TRIAL: NCT01865877
Title: Motor, Non-motor and Genetic Determinants of Progression and Complications in Parkinson's Disease: A Multicenter Cohort Study in Mexican Population (ReMePArk)
Brief Title: Motor, Non-motor and Genetic Determinants of Progression in Parkinson's Disease: A Mexican Multicenter Cohort Study
Acronym: ReMePARK
Status: Completed | Type: Observational
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Amin Cervantes-Arriaga, MD, MSc, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Other Study IDs: INNN 35/12; 182133 (Other Grant/Funding Number: CONACyT FOSSIS 182133)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Motor; Non-motor; Progression; Complications
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum and/or saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD Cohort: Subjects diagnosed with Parkinson's disease

SUMMARY:
The objective of the study is to assess the effect of motor, non-motor and genetic factors on the progression of Parkinson's disease as well as its impact on complications rates.

A large sample of Mexican subjects with Parkinson's disease attending several referral centers will be included.

Data collected will include disease severity and motor scales, non-motor scales as well as genotyping for monogenic forms of the disease.

Assessments will be performed every 6 months for two years.

DETAILED DESCRIPTION:
Demographic and clinical data will be collected after obtaining a signed informed consent.

Recruitment will be competitive. Data collected includes age, gender, motor phenotype, age at onset, age at diagnosis, smoking history, family history, antiparkinsonic treatment, other treatments and a complete neurological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease by the United Kingdom Parkinson's disease Society Brain Bank Criteria
* Any gender
* Any Hoehn and Yahr stage
* Written informed consent

Exclusion Criteria:

* Severe comorbidity that may limit proper neurological evaluation as judged by the investigator
* Subjects with atypical or secondary parkinsonism

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with idiopathic or genetic Parkinson's disease attending any of the participant sites in Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To assess motor scale change over time | Every 6 months for 2 years
  Motor symptoms will be assessed by proper and validated motor scales; also minimal clinically important change will be determined.

SECONDARY OUTCOMES:
To assess non-motor symptoms over time | Every 6 months for 2 years
  Non-motor symptoms will be assessed using proper validated scales. Frequency and severity will be recorded.
To assess quality of life change over time. | Every 6 months for 2 years
  Health-related quality of life will be assessed with proper validated clinimetric instruments.
To assess caregiver burden as disease progresses | Every 12 months for 2 years
  Caregiver burden will be assessed by proper validated scales.

OTHER OUTCOMES:
To assess the change in prevalence of neuropsychiatric symptoms over time | Every 12 months for 2 years
  Prevalence and incidence of depression, apathy, cognitive decline, psychosis and impulse control disorder will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Cervantes-Arriaga, MD,MSc, Principal Investigator — Instituto Nacional de Neurología y Neurocirugía
Locations (7):
- Mexico (7):
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital General de México, Mexico City, Mexico City
  - Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico City
  - Hospital Universitario, Monterrey, Nuevo León
  - Hospital Universitario, San Luis Potosí City, San Luis Potosí
  - Hospital Regional #1, Mérida, Yucatán
  - Hospital General de Zacatecas, Zacatecas City, Zacatecas

REFERENCES:
- [Result] Cervantes-Arriaga A, Rodriguez-Violante M, Lopez-Ruiz M, Estrada-Bellmann I, Zuniga-Ramirez C, Otero-Cerdeira E, Camacho-Ordonez A, Gonzalez-Latapi P, Morales-Briceno H, Martinez-Ramirez D. [Profile characterization of Parkinson's disease in Mexico: ReMePARK study]. Gac Med Mex. 2013 Sep-Oct;149(5):497-501. Spanish. PMID 24108335
- [Result] Cervantes Arriaga A, Rodriguez Violante M, Camacho Ordonez A, Gonzalez Latapi P, Lopez Ruiz M, Estrada Bellmann I, Zuniga Ramirez C, Otero Cerdeira E. [Time from motor symptoms onset to diagnosis of Parkinson's disease in Mexico]. Gac Med Mex. 2014 Dec;150 Suppl 2:242-7. Spanish. PMID 25643785
- See also: Instituto Nacional de Neurología y Neurocirugía — http://www.innn.salud.gob.mx